CLINICAL TRIAL: NCT06451185
Title: An Adaptive Randomised Controlled Trial, Performed in a Cardiothoracic Theatre and Critical Care Setting, to Investigate the Integrity and Durability of Standard Care Dressings Compared With Use of an Additional Haemostatic Powder, to Cover and Protect Central Venous Catheter Insertion Sites
Brief Title: Statseal® for Central Venous Catheter Insertion Sites in Critical Care
Acronym: SCENIC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Collaborators: Biolife LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 338511
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Central Line; Central Venous Catheter; Vascular Access; Critical Care; Hemostatic
Keywords: Adaptive; Randomized Controlled Trial; Low-intervention; Low-risk; Open Label; Pragmatic

STUDY DESIGN:
Intervention Model Description: A single centre, prospective, open label, randomised, controlled, adaptive investigation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Care Group (No Intervention): Following successful insertion of a central venous catheter into an internal jugular vein, the site will be covered with a standard care transparent dressing.
- Haemostatic Powder Group (Experimental): Following successful insertion of a central venous catheter into an internal jugular vein, the site will be covered with a haemostatic powder product beneath the standard care transparent dressing.
  Interventions: Other: A haemostatic mineral powder product.

INTERVENTIONS:
Other: A haemostatic mineral powder product. — The intervention is the addition of an approved and commercially available haemostatic powder product which is indicated for the temporary external control of bleeding. Recommended application is at central venous catheter insertion, prior to the site being covered with a transparent dressing. Comprising a hydrophilic polymer and potassium ferrate, once in contact with protein-rich body fluids, the mechanism of action of the powder is to dehydrate and to absorb exudate. This simultaneously forms a low pH seal barrier which is hostile to microbial penetration while also purporting to help maintain clean and dry environment beneath transparent site dressings.
  Arms: Haemostatic Powder Group

SUMMARY:
All participants in this clinical trial will be undergoing surgery and will have a central venous catheter (also known as a central line) placed in the large vein in the neck as part of their routine care.

The purpose of this clinical trial is to compare different ways of dressing central lines. In current standard care, central lines are stitched in place and covered with a protective transparent dressing. This standard care will be compared with the addition of a haemostatic powder beneath the transparent dressing. This powder product aids clotting at the level of the skin, meaning that it prevents or reduces bleeding while helping to maintain a dry and protected environment.

The main questions this clinical trial aims to answer are:

* Will the addition of a haemostatic powder increase the durability of central line dressings?
* What proportion of dressings required an unplanned change?
* The reason(s) for any unplanned change
* The incidence of bleeding around central line insertion sites
* Were any skin problems observed once the dressings were removed?

Once the dressings are applied, all central lines sites will be monitored as part of the participant's routine care. Participation in the clinical trial lasts as long as the first central line dressing remains in place. Central line dressings currently and routinely remain in place for up to, but not more than seven days. After this period, there will be no need for any research-related observations. Routine care will continue and will not be affected by the research. Participants will not be asked to make any extra visits over and above those needed for routine care.

DETAILED DESCRIPTION:
Current established practice recommends that central venous catheter (CVC) dressings that are clean dry and intact can safely remain in place for up to seven days. Bleeding and moisture at CVC insertion sites can lead to poor dressing adherence and to an environment favourable for microbial growth. Additional unplanned interactions are provoked such as undressing, cleaning and redressing the site; in some circumstances it may be necessary to change or to re-site the catheter. Each of these factors may increase the risk of infection while consuming additional healthcare time and resource.

The study will recruit patients undergoing surgery in a tertiary cardiothoracic hospital. Those selected will have planned CVC insertion. The majority of patients will have an increased bleeding risk due to the nature of cardiac surgery, usually requiring a number of agents to reduce their risk of thrombosis. Whilst there is a suitably individualised and patient-specific assessment of risk, the internal jugular is the preferred vein for a large proportion of our patients.

Haemostasis is the mechanism by which bleeding is stopped by the formation of a clot. In anticoagulated patients, clot formation is prolonged resulting in frequent oozing and bleeding around CVC insertion sites and to the soiling of dressings. Serous exudate, clammy skin and diaphoresis present additional challenges in this patient cohort. StatSeal® is an approved and commercially available haemostatic powder product indicated for the temporary external control of bleeding. Recommended application is at CVC insertion, prior to the site being covered with a transparent dressing. Comprising a hydrophilic polymer and potassium ferrate, once in contact with protein-rich body fluids, the mechanism of action of the powder is to dehydrate and to absorb exudate. This simultaneously forms a low pH seal barrier which is hostile to microbial penetration while also purporting to help maintain clean and dry environment beneath transparent dressings.

The objective of the study is to compare current standard care with use of an additional haemostatic powder.

Following the successful insertion of an internal jugular CVC in the theatre area, participants will be randomised in a 1:1 ratio into one of the following groups:

1. Current standard care group - where the site is covered with a transparent dressing.
2. Intervention group - where the powder will be applied around the CVC skin insertion site before being covered with the same transparent dressing.

This is a low-intervention, low-risk pragmatic study. The consent seeking process is proportionate and adapted to the design of the study.

Routine monitoring of each CVC site will follow. Each CVC insertion site will be observed from randomisation for a period of 168 hours (seven days) or up to the time of CVC removal or first dressing change (which ever event occurs soonest). The 7-day period has been selected as this would be the time of the first planned dressing change for the CVC placed at randomisation. Within this period, data will be collected to investigate the duration and integrity of each index dressing including the reasons for removal and, the skin status at removal.

Data collection will be electronic and will be performed by medical, nursing and other suitably qualified and trained staff thus facilitating multidisciplinary collaboration and integration of research with everyday clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Pre-Theatre Phase - Scheduled for insertion of an internal jugular CVC as part of their routine care

Theatre Phase

- Successful insertion of an internal jugular CVC

Exclusion Criteria:

Pre-Theatre phase

* Patients younger than 18 years of age
* Patients scheduled cannulation with more than one sheath or catheter into an ipsilateral internal jugular vein
* Patients with compromised skin integrity in the area to be covered with the CVC transparent dressing
* Patients who are scheduled to be transferred to another hospital at any time during the trial observation period of seven days post randomisation

Theatre phase

* Randomisation system not available
* Known allergy to study dressings
* Trial dressings not available
* Skin barrier product not available
* Securement suture not practicable
* The CVC insertion site cannot be covered with either a single conventional dressing or the haemostatic powder covered with a single transparent dressing
* Central line has a subcutaneous tunnel
* More than one ipsilateral central venous sheath or catheter in situ (or planned)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Time to first unplanned change of the index dressing. | Seven days
  Time to first unplanned change of the index dressing (measured in hours) from randomisation, or CVC removal (at any time) or planned index dressing removal (at seven days) - whichever is soonest.

SECONDARY OUTCOMES:
Reason(s) for an unplanned change of the index dressing | Seven days
  The reason(s) for an unplanned change of the index dressing
Proportion of index dressings that required an unplanned change | Seven days
  The proportion of index dressings that require an unplanned change in the period from randomisation to planned CVC removal or routinely scheduled dressing change
Skin status at dressing removal | Seven days
  Skin status at index dressing removal, defined as: erythema only, limited to ≤ 1.5cm of the CVC insertion site, and when extending >1.5cm up to and beyond the adhesive border of the transparent dressing and clinically assessed to be dressing-related. Evidence of mechanical skin injury suggested by rips or tears, with or without erythema extending up to 1.5cm beyond the adhesive border of the transparent dressing. Evidence of other skin disruption with or without erythema such as blisters or maceration within the same extended area of up to 1.5cm
Incidence of bleeding | Seven days
  The incidence of CVC insertion site related bleeding observed beneath the transparent portion of the dressing. As is best practice and standard care, all will prompt dressing change. Trial definition of bleeding: Grade 1 - dry blood observed in the vicinity of the puncture site, change of dressing (with usual site cleansing) being the only actions required. Note: blood that has formed a desiccated complex with the haemostatic powder is not considered contamination. Grade 2 - overt but minor bleeding requiring minimal bedside action(s) such as manual compression or application of wound adhesive. Grade 3 - continuous or significant overt bleeding requiring timely investigation such as ultrasound or radiological assessment, with action(s) informed by findings. Grade 4 - continuous or significant overt bleeding requiring urgent or emergency action

CONTACTS AND LOCATIONS:
Overall Officials: Rodney H Stables, MA DM BM BCh FRGS, Study Director — Liverpool Heart and Chest Hospital
Locations (1):
- Liverpool Heart and Chest Hospital NHS FoundationTrust, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data that underlie the results at publication will be made available on request.
Time Frame: For up to 24 months following publication.
Access Criteria: Prospective researchers should contact the Sponsor with details of their analysis plan and an assertion that they commit to open publication of their findings. Data will be provided without investigator support.
URL: https://www.lhch.nhs.uk